CLINICAL TRIAL: NCT00760500
Title: Surveillance of Influenza Virus Among Children With Febrile Respiratory Complaints Attending the Pediatric Clinic of the First Affiliated Hospital, Shantou University Medical College, Shantou, Guangdong, Mainland China
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: The University of Hong Kong (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: SIVFRC; N01AI70005 (NIH)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Influenza Type A; Influenza Type B

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal specimen taken by swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Nasopharyngeal Swab

INTERVENTIONS:
Other: Nasopharyngeal Swab — Nasopharyngeal Swab

SUMMARY:
The surveillance of influenza virus among children with febrile reparatory complaints attending the pediatric clinic in Shantou is an epidemiologic study to identify the type (influenza A or B) and the subtype of Influenza A of the isolates from children with febrile respiratory complaints who attend the pediatric clinic of the first Affiliated Hospital, Shantou University Medical College, Shantou Guangdong, China. Also this study investigates the genetic composition of all segments of isolated strains using standard molecular techniques and to make available the new strains of influenza viruses isolated from such children for the formulation of influenza vaccines. Clinical manifestation of the respiratory illness is recorded and single nasopharyngeal swab is obtained from eligible children. Viral culture is performed on the nasopharyngeal secretions. If influenza is isolated, this is characterized if it belongs to influenza A or B. If the virus is characterized as influenza A, further antigenic studies is done to determine subtype of influenza. Viral isolates is further studied to determine the genetic composition of the virus. Information obtained from the viral isolates is shared with the WHO and the CDC.

DETAILED DESCRIPTION:
OBJECTIVES

Primary objective:

* To identify the type (Influenza A or B) and the subtype of Influenza A of the isolates from children with febrile respiratory complaints who attend the pediatric clinic of the First Affiliated Hospital, Shantou University Medical College, Shantou, Guangdong, China.

Secondary objectives

* To investigate the genetic composition of all segments of isolated strains using standard molecular techniques.
* To make available the new strains of influenza viruses isolated from such children for the formulation of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0 day to 18 years.
* Patient was seen at the pediatric clinic of the First Affiliated Hospital within 7 days of the onset of signs and symptoms of febrile respiratory illness suspected to be of viral origin (temperature > 37.7ºC or reliable history of fever before being examined, and respiratory symptoms and signs such as cough, sore throat, and coryza).
* Parents agree to a nasopharyngeal specimen being taken by swab from their child.

Exclusion Criteria:

* Patient is too ill to tolerate a nasopharyngeal specimen swab.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the ages of 0 months and 18 years (inclusive) who have been seen at the pediatric clinic of the First Affiliated Hospital within 7 days of the onset of signs and symptoms of febrile respiratory illness suspected to be of viral origin (temperature > 37.7ºC or reliable history of fever before being examined, and respiratory symptoms and signs such as cough, sore throat, and coryza).
Sampling Method: Non-Probability Sample
Enrollment: 13201 (Actual)
Dates: Start 2004-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To identify Influenza A or B and the subtype of Influenza A of the isolates from children with febrile respiratory complaints who attend the pediatric clinic of the First Affiliated Hospital, Shantou University Medical College. | This is an epidemiologic study, there is no time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Miguela Caniza, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- First Affiliated Hospital, Shantou, Guangdong, China

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols